CLINICAL TRIAL: NCT03260452
Title: Comparison of Hematopoietic Stem Cell Activity in Adipose Tissue From Type 2 Diabetic Patients and Healthy Volunteers: Proof of Concept Study. White Adipose Tissue and Type 2 Diabetes Onset: WAT2DO
Brief Title: Comparison of Hematopoietic Stem Cell Activity in Adipose Tissue From Type 2 Diabetic Patients and Healthy Volunteers
Acronym: WAT2DO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/15/7739; 2017-A01697-46 (Other: ID-RCB)
Record Dates: First submitted 2017-07-27; First posted 2017-08-24 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-04

CONDITIONS: Type2 Diabetes
Keywords: Type 2 diabetes; Adipose tissue; Hematopoiesis; Inflammation; Macrophages
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation | interventions — Hematologic Tests

STUDY DESIGN:
Intervention Model Description: 20 male volunteers: 10 overweight/obese subjects with T2D and 10 healthy volunteers, age-matched.
  All volunteers will be treated in the same way.
Masking Description: All laboratory analyses will be performed blindly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): 'Abdominal subcutaneous biopsies and Blood test'
  Interventions: Procedure: Abdominal subcutaneous biopsies and Blood test

INTERVENTIONS:
Procedure: Abdominal subcutaneous biopsies and Blood test — Abdominal subcutaneous biopsies and blood test for each volunteer.

SUMMARY:
Based on solid preclinical results in mice and preliminary data in humans, this study aims to provide the proof of concept of the crucial role of the hematopoietic process occurring in human adipose tissue in the initiation of the inflammatory process at the origin of insulin resistance and type 2 diabetes (T2D). The main objective is to compare the number of pro-inflammatory macrophages derived from human adipose tissue hematopoietic stem cells (HSC) according to their origin, type 2 diabetes subjects or healthy volunteers.

DETAILED DESCRIPTION:
In mice, increasing data demonstrate a causal relationship between the inflammatory process in adipose tissue and the development of insulin resistance, resulting in type 2 diabetes occurrence. However, the mechanisms mediating inflammation and its metabolic consequences are still unclear. In humans, recent publications have suggested an important interaction between the metabolic status and medullar hematopoietic activity. A preliminary study performed by the STROMAlab's research team has identified functional hematopoietic stem cells in human adipose tissue samples, indicating that adipose tissue-hematopoiesis is an active mechanism.

To determine whether an alteration in adipose tissue-hematopoiesis could be a hallmark of type 2 diabetes in human, biopsies of subcutaneous adipose tissue will be performed in 2 groups of 10 volunteers: overweight/obese type 2 diabetes subjects versus healthy volunteers, matched on age.

Then, hematopoietic stem cells extracted from human biopsies will be grafted into immunodeficient mice and after 12 weeks, flow cytometry using antibodies specific for human cell surface markers will be performed to quantify proinflammatory macrophages derived from human adipose tissue-hematopoietic stem cells.

ELIGIBILITY:
Inclusion Criteria:

* No major weight variation for at least 3 months
* Biological assessment without clinically significant anomaly from the point of view of the investigator.
* Acceptance of constraints related to participation in the study
* Acceptance of participation in the constitution of a cell bank, a tissue bank and a serum library.
* Affiliation to a social security scheme.

Type 2 diabetic subjects:

* Type 2 diabetes (discovered after the age of 35 years, without inaugural ketosis and absence of insulin therapy during the first year).
* 40 to 60 year-old.
* BMI between 27 and 35 kg / m² (included).
* Treated by modification of lifestyle alone or associated to oral anti-diabetic therapy only.
* With stable oral anti-diabetic treatment for at least 3 months.
* HbA1c ≤ 8.5%.

Healthy Volunteers:

* BMI between 23 and 27 kg / m² (included).
* 37 to 63 year-old, age-matched to a type 2 diabetes subject ± 5 years.
* Fasting blood glucose < 1,10 g / L.
* HbA1c within normal limits (4 to 6%).

Exclusion Criteria:

* Excessive chronic alcohol consumption (> 30 g / day or 210 g / week).
* Tobacco consumption> 10 cigarettes / day that cannot be stopped for 24 hours.
* Anti-diabetic treatments that require sub-cutaneous injections
* History of chronic or acute hematological pathology.
* Systemic or acute inflammatory pathology.
* Treatment with antiplatelet agents, non-steroidal anti-inflammatory drugs, glucocorticoids (excluding eye drops and sprays), or other immunosuppressive drugs.
* History of cancer (except basal cell carcinoma).
* Allergy to xylocaine or one of its derivatives.
* Any significant pathology at the discretion of the investigator.
* Any biological anomaly at the discretion of the investigator.
* Positive human immunodeficiency virus serology.
* Positive hepatitis B serology.
* Positive hepatitis C serology.
* Glomerular filtration rate less than 60 ml / min
* Aspartate aminotransferase or alanine aminotransferase higher than 2.5-fold the upper normal value.
* Hypertriglyceridemia > 2.5 g / l
* Person under the protection of justice, guardianship or curators.
* Subject involved in another research protocol or in an exclusion period from another research protocol.
* Cognitive disorder or mental pathology (at the discretion of the investigator).

Ages: 37 Years to 63 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-01-24 (Actual)

PRIMARY OUTCOMES:
Number of pro-inflammatory macrophages derived from human adipose tissue in mice transplanted with adipose tissue-hematopoietic stem cells . | Day 3 - Day 45
  The investigators expect that the number of pro-inflammatory macrophages derived from human adipose tissue will be significantly higher in mice transplanted with adipose tissue-hematopoietic stem cells isolated from diabetic subjects compared to those from healthy volunteers.

SECONDARY OUTCOMES:
Comparison of hematopoietic activity in vitro between both groups of subjects. | Day 3 - Day 45
  Evaluated by flow cytometry.
Comparison of the number of the other cell types derived from the human adipose tissue-hematopoietic stem cells between both groups of grafted mice. | Day 3 - Day 45
  Evaluated by flow cytometry.
Comparison of the phenotype of the other cell types derived from the human adipose tissue-hematopoietic stem cells between both groups of grafted mice. | Day 3 - Day 45
  Evaluated by flow cytometry.
Comparison of the expression of genes coding for human inflammatory molecules in the adipose tissue of transplanted mice. | Day 3 - Day 45
  Evaluated by Real-Time Quantitative Reverse Transcription Polymerase Chain Reaction. Main parameters analysed : Interleukin-6, Interleukin-1béta, Plasminogen activator inhibitor-1, Monocyte Chemoattractant Protein-1.
Comparison of the metabolic profile of the transplanted mice evaluated by the grafted mice's glycemia. | Day 3 - Day 45
  According to the origin of the grafted hematopoietic stem cells (diabetic or healthy voluntary subjects).
Comparison of the metabolic profile of the transplanted mice evaluated by the grafted mice's insulinemia. | Day 3 - Day 45
  According to the origin of the grafted hematopoietic stem cells (diabetic or healthy voluntary subjects).
Comparison of the metabolic profile of the transplanted mice evaluated by the grafted mice's oral glucose tolerance test. | Day 3 - Day 45
  According to the origin of the grafted hematopoietic stem cells (diabetic or healthy voluntary subjects).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre GOURDY, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse - Rangueil, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Casteilla L, Planat-Benard V, Laharrague P, Cousin B. Adipose-derived stromal cells: Their identity and uses in clinical trials, an update. World J Stem Cells. 2011 Apr 26;3(4):25-33. doi: 10.4252/wjsc.v3.i4.25. PMID 21607134
- [Background] Bour S, Caspar-Bauguil S, Iffiu-Soltesz Z, Nibbelink M, Cousin B, Miiluniemi M, Salmi M, Stolen C, Jalkanen S, Casteilla L, Penicaud L, Valet P, Carpene C. Semicarbazide-sensitive amine oxidase/vascular adhesion protein-1 deficiency reduces leukocyte infiltration into adipose tissue and favors fat deposition. Am J Pathol. 2009 Mar;174(3):1075-83. doi: 10.2353/ajpath.2009.080612. Epub 2009 Feb 13. PMID 19218346
- [Background] Brooks-Worrell B, Narla R, Palmer JP. Biomarkers and immune-modulating therapies for type 2 diabetes. Trends Immunol. 2012 Nov;33(11):546-53. doi: 10.1016/j.it.2012.07.002. Epub 2012 Aug 14. PMID 22897868
- [Background] Cancello R, Clement K. Is obesity an inflammatory illness? Role of low-grade inflammation and macrophage infiltration in human white adipose tissue. BJOG. 2006 Oct;113(10):1141-7. doi: 10.1111/j.1471-0528.2006.01004.x. Epub 2006 Aug 10. PMID 16903845
- [Background] Caspar-Bauguil S, Cousin B, Bour S, Casteilla L, Penicaud L, Carpene C. Adipose tissue lymphocytes: types and roles. J Physiol Biochem. 2009 Dec;65(4):423-36. doi: 10.1007/BF03185938. PMID 20358356
- [Background] Cousin B, Andre M, Arnaud E, Penicaud L, Casteilla L. Reconstitution of lethally irradiated mice by cells isolated from adipose tissue. Biochem Biophys Res Commun. 2003 Feb 21;301(4):1016-22. doi: 10.1016/s0006-291x(03)00061-5. PMID 12589814
- [Background] Dalmas E, Tordjman J, Guerre-Millo M, Clement K. [Adipose tissue, a new playground for immune cells]. Med Sci (Paris). 2011 Nov;27(11):993-9. doi: 10.1051/medsci/20112711016. Epub 2011 Nov 30. French. PMID 22130027
- [Background] Han J, Koh YJ, Moon HR, Ryoo HG, Cho CH, Kim I, Koh GY. Adipose tissue is an extramedullary reservoir for functional hematopoietic stem and progenitor cells. Blood. 2010 Feb 4;115(5):957-64. doi: 10.1182/blood-2009-05-219923. Epub 2009 Nov 6. PMID 19897586
- [Background] Nagareddy PR, Murphy AJ, Stirzaker RA, Hu Y, Yu S, Miller RG, Ramkhelawon B, Distel E, Westerterp M, Huang LS, Schmidt AM, Orchard TJ, Fisher EA, Tall AR, Goldberg IJ. Hyperglycemia promotes myelopoiesis and impairs the resolution of atherosclerosis. Cell Metab. 2013 May 7;17(5):695-708. doi: 10.1016/j.cmet.2013.04.001. PMID 23663738
- [Background] Nikolajczyk BS, Jagannathan-Bogdan M, Denis GV. The outliers become a stampede as immunometabolism reaches a tipping point. Immunol Rev. 2012 Sep;249(1):253-75. doi: 10.1111/j.1600-065X.2012.01142.x. PMID 22889227
- [Background] Poglio S, De Toni-Costes F, Arnaud E, Laharrague P, Espinosa E, Casteilla L, Cousin B. Adipose tissue as a dedicated reservoir of functional mast cell progenitors. Stem Cells. 2010 Nov;28(11):2065-72. doi: 10.1002/stem.523. PMID 20845475
- [Background] Poglio S, De Toni F, Lewandowski D, Minot A, Arnaud E, Barroca V, Laharrague P, Casteilla L, Cousin B. In situ production of innate immune cells in murine white adipose tissue. Blood. 2012 Dec 13;120(25):4952-62. doi: 10.1182/blood-2012-01-406959. Epub 2012 Oct 15. PMID 23071275
- [Background] Prunet-Marcassus B, Cousin B, Caton D, Andre M, Penicaud L, Casteilla L. From heterogeneity to plasticity in adipose tissues: site-specific differences. Exp Cell Res. 2006 Apr 1;312(6):727-36. doi: 10.1016/j.yexcr.2005.11.021. Epub 2005 Dec 28. PMID 16386732
- [Background] Richardson VR, Smith KA, Carter AM. Adipose tissue inflammation: feeding the development of type 2 diabetes mellitus. Immunobiology. 2013 Dec;218(12):1497-504. doi: 10.1016/j.imbio.2013.05.002. Epub 2013 May 16. PMID 23816302
- [Background] Shapiro H, Lutaty A, Ariel A. Macrophages, meta-inflammation, and immuno-metabolism. ScientificWorldJournal. 2011;11:2509-29. doi: 10.1100/2011/397971. Epub 2011 Dec 28. PMID 22235182
- [Background] Spinetti G, Cordella D, Fortunato O, Sangalli E, Losa S, Gotti A, Carnelli F, Rosa F, Riboldi S, Sessa F, Avolio E, Beltrami AP, Emanueli C, Madeddu P. Global remodeling of the vascular stem cell niche in bone marrow of diabetic patients: implication of the microRNA-155/FOXO3a signaling pathway. Circ Res. 2013 Feb 1;112(3):510-22. doi: 10.1161/CIRCRESAHA.112.300598. Epub 2012 Dec 18. PMID 23250986
- [Background] Weisberg SP, McCann D, Desai M, Rosenbaum M, Leibel RL, Ferrante AW Jr. Obesity is associated with macrophage accumulation in adipose tissue. J Clin Invest. 2003 Dec;112(12):1796-808. doi: 10.1172/JCI19246. PMID 14679176
- [Background] Xu H, Barnes GT, Yang Q, Tan G, Yang D, Chou CJ, Sole J, Nichols A, Ross JS, Tartaglia LA, Chen H. Chronic inflammation in fat plays a crucial role in the development of obesity-related insulin resistance. J Clin Invest. 2003 Dec;112(12):1821-30. doi: 10.1172/JCI19451. PMID 14679177
- [Background] Ito R, Takahashi T, Katano I, Ito M. Current advances in humanized mouse models. Cell Mol Immunol. 2012 May;9(3):208-14. doi: 10.1038/cmi.2012.2. Epub 2012 Feb 13. PMID 22327211